CLINICAL TRIAL: NCT03938337
Title: Clinical Trial of Abemaciclib in Combination With Pembrolizumab in Patients With Metastatic or Recurrent Head and Neck Cancer
Brief Title: Abemaciclib and Pembrolizumab in Metastatic or Recurrent Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated study due to higher incidence of pulmonary toxicity than expected, including death
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Eddy Yang, Primary Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAB 1891
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Head and Neck Cancer
Keywords: immunotherapy; abemaciclib; pembrolizumab; Cyclin-Dependent Kinase (CDK): CDK4; Cyclin-Dependent Kinase (CDK): CDK6
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 Not Previously Treated (Experimental): Patients with metastatic or recurrent head and neck cancer who have not been treated previously with immunotherapy.
  Interventions: Drug: Cohort 1 Not Previously Treated
- Cohort 2 Treated Previously (Experimental): Patients with metastatic or recurrent head and neck cancer who have been treated previously with immunotherapy.
  Interventions: Drug: Cohort 2 Treated Previously

INTERVENTIONS:
Drug: Cohort 1 Not Previously Treated — Abemaciclib 150mg by mouth twice daily Pembrolizumab 200mg IV every 3 weeks
  Other Names: CDK4:CDK6
  Arms: Cohort 1 Not Previously Treated
Drug: Cohort 2 Treated Previously — Abemaciclib 150mg by mouth twice daily Pembrolizumab 200mg IV every 3 weeks
  Other Names: CDK4:CDK6
  Arms: Cohort 2 Treated Previously

SUMMARY:
To assess the objective response rate of tumor lesions to abemaciclib in combination with pembrolizumab in patients with metastatic or recurrent squamous cell carcinoma of head and neck.

DETAILED DESCRIPTION:
Immunotherapy has been recently approved for patients with metastatic or recurrent squamous cell carcinoma of the head and neck. However, only a small percentage of patients experience long-term control, necessitating new therapeutic strategies. Recently, it was shown preclinically and in breast tumors that abemaciclib stimulates production of type III interferons and hence enhances tumor antigen presentation. Abemaciclib also suppressed the proliferation of regulatory T cells. These events promote cytotoxic T-cell-mediated clearance of tumor cells, which is further enhanced by the addition of immune checkpoint blockade. Based on these data, a phase II trial in patients with metastatic or recurrent head and neck cancer who are eligible for immunotherapy is proposed to investigate the combination of abemaciclib with pembrolizumab. Tumor & blood analysis for interferon gamma signature will be explored as possible biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed (core biopsy proven) metastatic or recurrent squamous cell carcinoma of head and neck
* Adequate pulmonary and cardiac function
* Available archived tissue of primary tumor or resected tumor specimen with adequate samples
* Prior treatment with immune checkpoint inhibitor is not allowed in cohort 1 patients. Patients in cohort 2 should have failed or progressed on prior immune checkpoint inhibitor
* Eastern Cooperative Oncology Group Performance Status(ECOG PS) = 0 or 1
* Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse [CTCAE] Grade <= 1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization. A washout period of at lease 21 days is required between last chemotherapy dose and randomization (provided the patient did not receive radiotherapy)
* Patients who received adjuvant radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization
* The patient is able to swallow oral medications
* Adequate hematologic and end-organ function
* Absolute Neutrophil Count (ANC) >= 1500/mm3
* Platelet count ≥ 100,000/mm3
* Hemoglobin (Hb) ≥ 8g/dl (Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion)
* Creatinine (Cr) ≤ 1.5 x Upper Limit of Normal (ULN) or Creatinine Clearance (CrCl) ≥ 60 ml/min
* Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert syndrome, who can have total Bilirubin < 2.0 x ULN and direct bilirubin within normal limits are permitted.)
* Aspartate Aminotransferase (AST) and Alanine aminotransferase (ALT) and alkaline phosphatase ≤ ULN
* Agreement to remain abstinent or use appropriate contraception, among women of childbearing potential
* Willingness and ability to consent for self to participate in study
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Autoimmune disease (Note: Vitiligo, type 1 diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, and conditions not expected to recur in the absence of an external trigger are permitted.)
* Condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to study treatment (Note: Inhaled and topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.)
* Preexisting medical condition(s) that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Immunosuppression, of any kind
* Prior treatment with Cyclin-Dependent Kinase(CDK) 4/6 Inhibitor
* Major surgical procedure or significant traumatic injury within 4 weeks prior to study treatment, and must have fully recovered from any such procedure
* Personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest
* Angina, myocardial infarction (MI), symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack TIA), arterial embolism, pulmonary embolism, percutaneous transluminal coronary angioplasty (PTCA), or coronary artery bypass grafting (CABG) within 6 months prior to study treatment
* Known active viral or non-viral hepatitis or cirrhosis
* Any active infection requiring systemic treatment, positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA).
* History of gastrointestinal perforation or fistula in the 6 months prior to study treatment, unless underlying risk has been resolved (e.g., through surgical resection or repair)
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
* Pregnancy or breastfeeding - Female patients must be surgically sterile (i.e., ≥6 weeks following surgical bilateral oophorectomy with or without hysterectomy or tubal ligation) or be postmenopausal, or must agree to use effective contraception during the study and for 4 months following last dose of treatment. All female patients of reproductive potential must have a negative pregnancy test (serum or urine) within 7 days prior to study treatment. Male patients must be surgically sterile or must agree to use effective contraception during the study and for 4 months following last dose of treatment.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Yang, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
To Be Determined
Supporting Information: Study Protocol, SAP, ICF
Time Frame: As long as study record is posted on CT.gov
Access Criteria: To Be Determined

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: study terminated prematurely due to toxicity from other trials with this combination
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Objective Response Rate of Tumor Lesions Using Scans
Description: Patients will be evaluated for their tumor response to treatment using RECIST criteria on their scans
Time Frame: Baseline
Population: No analysis was performed since study terminated prematurely due to toxicity from other trials with this combination
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: To Assess the Objective Response Rate of Tumor Lesions Using Scans
Description: Patients will be evaluated for their tumor response to treatment using RECIST criteria on their scans
Time Frame: Baseline to 5 months
Population: No analysis was performed since study terminated prematurely due to toxicity from other trials with this combination
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: To Assess the Objective Response Rate of Tumor Lesions Using Scans
Description: Patients will be evaluated for their tumor response to treatment using RECIST criteria on their scans
Time Frame: Baseline to 8 months
Population: No analysis was performed since study terminated prematurely due to toxicity from other trials with this combination
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants Experiencing Adverse Events Grade 3 or Greater
Description: Measure adverse events grade 3 or greater to evaluate safety and tolerability
Time Frame: Baseline to 1 month
Population: No analysis was performed since study terminated prematurely due to toxicity from other trials with this combination
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants Experiencing Adverse Events Grade 3 or Greater
Description: Measure adverse events grade 3 or greater to evaluate safety and tolerability
Time Frame: Baseline to 6 months
Population: No analysis was performed since study terminated prematurely due to toxicity from other trials with this combination
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants Experiencing Adverse Events Grade 3 or Greater
Description: Measure adverse events grade 3 or greater to evaluate safety and tolerability
Time Frame: Baseline to 12 months
Population: No analysis was performed since study terminated prematurely due to toxicity from other trials with this combination
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: To Assess Progression Free Survival (PFS)
Description: Using scan results to assess whether tumor has progressed and the time;
Time Frame: baseline to 6 months
Population: No analysis was performed since study terminated prematurely due to toxicity from other trials with this combination
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: To Assess Progression Free Survival (PFS)
Description: Using scan results to assess whether tumor has progressed and the time;
Time Frame: baseline to 12 months
Population: No analysis was performed since study terminated prematurely due to toxicity from other trials with this combination
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: To Assess Overall Survival
Description: time that the patient is experiencing survival
Time Frame: baseline to 6 months
Population: No analysis was performed since study terminated prematurely due to toxicity from other trials with this combination
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: To Assess Overall Survival
Description: time that the patient is experiencing survival
Time Frame: baseline to 12 months
Population: No analysis was performed since study terminated prematurely due to toxicity from other trials with this combination
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: To Assess the Time to Tumor Response
Description: using scan results to assess the time it takes for the tumor to respond to treatment
Time Frame: baseline to 6 months
Population: No analysis was performed since study terminated prematurely due to toxicity from other trials with this combination
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: To Assess the Time to Tumor Response
Description: using scan results to assess the time it takes for the tumor to respond to treatment
Time Frame: baseline to 12 months
Population: No analysis was performed since study terminated prematurely due to toxicity from other trials with this combination
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: To Assess the Duration of Response
Description: using scan results to measure the total amount of time that the tumor is responding to treatment
Time Frame: baseline to 6 months
Population: No analysis was performed since study terminated prematurely due to toxicity from other trials with this combination
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: To Assess the Duration of Response
Description: using scan results to measure the total amount of time that the tumor is responding to treatment
Time Frame: baseline to 12 months
Population: No analysis was performed since study terminated prematurely due to toxicity from other trials with this combination
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline through 8 months
Description: Since study terminated prematurely due to toxicity from other trials with this combination, there were no SAEs and no mortality observed
Arm/Group | Cohort 1 Not Previously Treated | Cohort 2 Treated Previously
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Not Previously Treated (N=1) | Cohort 2 Treated Previously (N=0)
Afebrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | NA
Creatinine Increased (Renal and urinary disorders) | 1 (1) | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | NA
Fatigue (General disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT03938337/Prot_SAP_000.pdf